CLINICAL TRIAL: NCT06268067
Title: The Association of Kidney Uptake at F-18 FDG PET/CT Studies and Renal Function Status
Brief Title: Kidney Uptake at F-18 FDG PET/CT Studies and Renal Function Status
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana Mahmoud Farghali, Rana Mahmoud Farghali, Assiut University
Other Study IDs: Renal uptake at F18 FDG PET/CT
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Renal Uptake at F-18-FDG PET/CT
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic kidney diseased patiens: chronic kidney diseased patients
  Interventions: Device: PET/CT
- Normal: normal subjects
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT — F-18 FDG PET/CT studies

SUMMARY:
Searching for a possible correlation between renal uptake at F-18-FDG PET/CT and renal functional parameters in both normal subjects and patients with CKD.

DETAILED DESCRIPTION:
F-18-Fluoro-Deoxy-Glucose Positron Emission Tomography (F-18 FDG PET/CT) is a hybrid imaging modality that in the last few years has been gaining more attention, due to its ability for evaluation different conditions, both neoplastic or benign. In the urinary tract, FDG is filtered by the glomerulus and is not reabsorbed by the renal tubules. So, significant activity may be displayed in any part of the urinary tract. Chronic kidney disease is highly prevalent and associated with higher cardiovascular risk. CKD is diagnosed when an estimated glomerular filtration rate (EGFR) lower than 60 mL/min/1.73 m2 present for at least three months or by alteration in the renal structure[3]. The Kidney Disease: Improving Global Outcomes (KDIGO) CKD guidelines recommend use of the EGFR for determination of the disease because of its simplicity, cost-effectiveness, and accuracy in predicting renal function in standard conditions. The estimating equation for the assessment of EGFR in adults is the CKD Epidemiology Collaboration (CKD-EPI).

In some cases, it has been reported that the impairment of renal function doesn't significantly compromise the clearance of background activity of F-18-FDG. In contrast, other papers observed that CKD patients have a higher physiological tracer uptake in the liver and blood pool. Different studies investigated the ability of CKD in modification of the F-18-FDG uptake during a PET/CT scan have also been published with contradictory results.

Therefore, we search for the association between renal uptake at F-18-FDG PET/CT and renal functional parameters in both normal subjects and CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing PET/CT examination for oncologic or non-oncologic purposes.

Exclusion Criteria:

* Patients underwent PET/CT examination with age under 18 years.
* Presence of pathological conditions affecting kidneys (e.g., cancers, inflammation, polycystic kidney disease)
* Inability to stay still for the duration of the scan.
* Claustrophobia.
* Patients with uncontrolled diabetics (blood glucose >200 mg/dl immediately before PET/CT scan)
* Pregnant females.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing PET/CT examination for oncologic or non-oncologic purposes.
  For all the patients included in this study, data about serum Cr levels and estimated glomerular filtration rate (EGFR) calculated with the CKD-EPI formula.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
significance of renal uptake at F18-FDG PET CT studies | one year
  The study assesses the significance of renal uptake at F18-FDG PET CT studies as regards Cr levels and EGFR.

SECONDARY OUTCOMES:
Early detection of patients with CKD | one year
  • Early detection of patients with CKD to initiate appropriate treatment for them, with subsequently improving the survival and quality of life.

REFERENCES:
- [Result] Dondi F, Pisani AR, Lucarelli NM, Gazzilli M, Talin A, Albano D, Rubini D, Maggialetti N, Rubini G, Bertagna F. Correlation between Kidney Uptake at [18F]FDG PET/CT and Renal Function. J Pers Med. 2023 Dec 28;14(1):40. doi: 10.3390/jpm14010040. PMID 38248741
- [Result] Ammirati AL. Chronic Kidney Disease. Rev Assoc Med Bras (1992). 2020 Jan 13;66Suppl 1(Suppl 1):s03-s09. doi: 10.1590/1806-9282.66.S1.3. PMID 31939529